CLINICAL TRIAL: NCT03203668
Title: Diagnostic Value of 18F-fluorocholine PET/CT Imaging in Localization of Hyperfunctioning Parathyroid Tissue in Hyperparathyroidism
Brief Title: 18F-fluorocholine PET/CT Imaging in Hyperparathyroidism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Institute of Oncology Ljubljana (Other)
Responsible Party: Principal Investigator, Luka Lezaic MD PhD, MD PhD, University Medical Centre Ljubljana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 77/11/12
Record Dates: First submitted 2017-04-17; First posted 2017-06-29 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Hyperparathyroidism
Keywords: Hyperparathyroidism; Imaging; Scintigraphy; 18F-choline; 18F-fluorocholine; PET; PET/CT
MeSH Terms: conditions — Hyperparathyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Choline PET/CT (Other): Choline PET/CT imaging added to conventional imaging assessment in hyperparathyroidism (parathyroid scintigraphy, ultrasound, CT or MRI if indicated)
  Interventions: Radiation: 18F-choline PET/CT

INTERVENTIONS:
Radiation: 18F-choline PET/CT — 18F-choline PET/CT imaging (neck, mediastinum)

SUMMARY:
To assess the efficiency of 18F-fluorocholine PET/CT in localization of hyperfunctioning parathyroid tissue in hyperparathyroidism, thereby enabling minimally invasive surgical approaches with fewer complications and comparable success rates

DETAILED DESCRIPTION:
Primary hyperparathyroidism is a common endocrine disorder for which the diagnosis is biochemical and therapy surgical in the vast majority of cases; in secondary and tertiary hyperparathyroidism, surgical treatment is usually chosen when conservative measures fail to control the condition. The previously used surgical approach of bilateral neck exploration is being replaced by minimally invasive procedures, whose advantage is shorter duration of operation and general anesthesia, lower morbidity and fewer complications with comparable success rates.

A prerequisite for minimally invasive surgery is successful localization of the offending parathyroid tissue. Most commonly used imaging modality for this purpose is parathyroid scintigraphy with 99mTc-sestaMIBI, usually supplemented by ultrasound of the neck. Overall, parathyroid scintigraphy is a sensitive method for localization of hyperfunctioning parathyroid tissue; however, its diagnostic performance is significantly lower in patients with multiple parathyroid lesions.

In comparison to conventional nuclear medicine imaging approaches for localization of the offending parathyroid tissue, positron emission tomography with computed tomography (PET/CT) offers superior image resolution with an additional advantage of attenuation correction and co-registration of functional and anatomical information. 18F-fluorocholine is a PET tracer which is commonly used for prostate cancer imaging. In contrast to 18F-fluorodeoxyglucose (18F-FDG), it is also taken up by well-differentiated neoplasms in which 18F-FDG uptake is unreliable. The investigators hypothesize that 18F-fluorocholine might be efficiently taken up by parathyroid adenomata and/or hyperplasia.

The aim of this study is to investigate the efficiency of localization of hyperfunctioning parathyroid tissue with 18F-fluorocholine PET/CT in patients with primary hyperparathyroidism and to compare its efficiency to conventional scintigraphic imaging methods for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Biochemically proven hyperparathyroidism (elevated iPTH, elevated on normal Ca2+) or elevated Ca2+ and inadequately supressed iPTH

Exclusion Criteria:

* Age under 18 years
* Pregnancy
* Clinical history of oncological, inflammatory/infectious disease of the head and neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity & Specificity | 3 months
  Ability to detect the hyperfunctioning parathyroid tissue

SECONDARY OUTCOMES:
Biochemical/clinical outcome - iPTH levels | 1 year
  Normalization of biochemical abnormalities related to hyperfunctioning parathyroid tissue (iPTH levels [pg/mL])
Biochemical/clinical outcome - Ca2+ levels | 1 year
  Normalization of biochemical abnormalities related to hyperfunctioning parathyroid tissue (Ca2+ levels [mmol/L])
Improvement in patient management - operating time | 3 years
  Duration of surgical procedure (minutes)
Improvement in patient management - duration of hospital stay | 3 years
  Duration of hospital stay (hours)
Improvement in patient management - complications of surgery | 3 years
  Complications (number)
Improvement in patient management - cost | 3 years
  Expenses of surgical/hospital management (EUR)

CONTACTS AND LOCATIONS:
Locations (1):
- Department for nuclear medicine, University medical centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lezaic L, Rep S, Sever MJ, Kocjan T, Hocevar M, Fettich J. (1)(8)F-Fluorocholine PET/CT for localization of hyperfunctioning parathyroid tissue in primary hyperparathyroidism: a pilot study. Eur J Nucl Med Mol Imaging. 2014 Nov;41(11):2083-9. doi: 10.1007/s00259-014-2837-0. Epub 2014 Jul 26. PMID 25063039
- [Result] Rep S, Lezaic L, Kocjan T, Pfeifer M, Sever MJ, Simoncic U, Tomse P, Hocevar M. Optimal scan time for evaluation of parathyroid adenoma with [(18)F]-fluorocholine PET/CT. Radiol Oncol. 2015 Nov 27;49(4):327-33. doi: 10.1515/raon-2015-0016. eCollection 2015 Dec. PMID 26834518
- [Result] Hocevar M, Lezaic L, Rep S, Zaletel K, Kocjan T, Sever MJ, Zgajnar J, Peric B. Focused parathyroidectomy without intraoperative parathormone testing is safe after pre-operative localization with 18F-Fluorocholine PET/CT. Eur J Surg Oncol. 2017 Jan;43(1):133-137. doi: 10.1016/j.ejso.2016.09.016. Epub 2016 Oct 21. PMID 27776943